CLINICAL TRIAL: NCT05606081
Title: Predicting Risk for Post-polypectomy Colorectal Cancer
Acronym: PREDICT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Alternative method of implementation, study not needed
Sponsor: Kaiser Permanente (Other)
Collaborators: The Permanente Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1547728-4
Record Dates: First submitted 2022-10-07; First posted 2022-11-04 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Neoplasm, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The risk prediction model is being applied to patients who are awaiting surveillance colonoscopy at select KPNC service areas to help identify those at highest risk for colorectal cancer based on their risk scores. The prediction model is being used in 2-3 service area to identify about 60-80 patients per month who are at highest risk for colorectal cancer based on their risk scores. Risk scores represent one of a number of factors being considered for prioritizing patients for colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Use of risk prediction scores (Experimental): The prediction model is being used to identify patients who are at highest risk for colorectal cancer based on their risk scores.
  Interventions: Device: Logistic regression risk model

INTERVENTIONS:
Device: Logistic regression risk model — Logistic regression model to assign risk score, plus time overdue and PROMPT risk category

SUMMARY:
This originated as an observational study of Kaiser Permanente Northern California (KPNC) patients with a history of adenoma diagnosed by colonoscopy who received a subsequent surveillance colonoscopy between 2014 and 2019. The original goal of the study was to develop a risk prediction model that would help identify patients at highest risk for a diagnosis of advanced neoplasia (colorectal cancer and/or advanced adenoma) at or within 6 months following their surveillance colonoscopy. Candidate predictors of interest included patient demographics, medical history, and details related to the index colonoscopy. The investigators are now at the implementation stage and applying the risk prediction model to patients awaiting surveillance colonoscopy at select KPNC service areas to help identify those at highest risk for colorectal cancer based on their risk scores.

DETAILED DESCRIPTION:
In the implementation stage, the risk prediction model is being applied to patients who are awaiting surveillance colonoscopy at select KPNC service areas to help identify those at highest risk for colorectal cancer based on their risk scores. The prediction model is being used in 2-3 service area to identify about 60-80 patients per month who are at highest risk for colorectal cancer based on their risk scores. Risk scores represent one of a number of factors being considered for prioritizing patients for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients are on the current colonoscopy pending list; excluding those who were fecal immunochemical test-positive, screening colonoscopies, had a colonoscopy in last 12 months or on a voluntary "pause" list

* Hereditary colorectal cancer syndrome (e.g. Lynch syndrome)
* Diagnostic, fecal immunochemical test -positive, or screening indication for colonoscopy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of colorectal neoplasia per number of colonoscopies performed | 1 year
  The investigators anticipate observing changed rates of colorectal neoplasia per number of colonoscopies performed on account of prioritizing higher risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Levin, MD, Principal Investigator — Kaiser Permanente Northern California, Division of Research
Locations (1):
- Kaiser Permanente Northern California Division of Research, Oakland, California, United States